CLINICAL TRIAL: NCT03096509
Title: MISSION ABC: Modern Innovative Solutions to Improve Outcomes in Asthma, Breathlessness and COPD - Participatory Action Research to Evaluate the Delivery of the MISSION ABC Service Model and Assess Health Service and Clinical Outcomes
Brief Title: Participatory Action Research to Evaluate the Delivery of the MISSION ABC Service Model and Assess Health Service and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Wessex Academic Health Science Network (Unknown); East Hampshire Better Local Care Fund (Unknown); Pfizer (Industry); The Health Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2016/84
Record Dates: First submitted 2017-03-01; First posted 2017-03-30 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: COPD; Asthma; Breathlessness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MISSION ABC Integrated Care clinic — The Investigators have developed a model of care incorporating key innovations for patients with asthma, COPD and undifferentiated breathlessness. This service is being implemented within Wessex CCGs.

SUMMARY:
Innovations aimed at improving new patient identification, diagnosis, nonpharmacological treatment, supported self-management, and remote monitoring, together with new methods of clinical support could improve outcomes in patients with respiratory disease. The Investigators have developed a model of care incorporating key innovations for patients with asthma, COPD and undifferentiated breathlessness. This service is being implemented within Wessex CCGs. The investigators will assess whether the implementation of the service is effective, and how it can be adjusted, in addition to introducing innovations to assess whether the expected benefits for patients are realised.

DETAILED DESCRIPTION:
A combination of study designs are required to evaluate all aspects of the service:

* Participatory action research approach, involving real-time evaluation at each clinic to inform subsequent clinics
* Before-and-after study for patient outcomes pre-clinic attendance and post-clinic attendance.
* Qualitative methods (interviews, focus groups)

Evaluation of the clinic cycles will include consideration of qualitative data from patients, carers and healthcare professionals, in addition to quantitative outcomes for service implementation and patient factors (i.e. uptake of the service and benefits realised in-session), including those in the following areas:

* Clinic process
* Education and supported self-management
* Added value of diagnostic tools (new diagnoses)
* Applicability and use of treatment tools and treatment tailoring
* Self-monitoring appropriateness and uptake
* Balance measures (e.g. increased secondary care traffic)

The longer-term impact of the service will be evaluated using clinical and health service outcomes such as:

* Hospitalisations for airways disease
* perceived disease control (symptom scores etc)
* exacerbation frequency
* health-related quality of life
* Patient Activation Measures (PAM)
* Treatments used
* Healthcare resource use (primary and secondary care)

ELIGIBILITY:
Inclusion Criteria:

* Attendance at a MISSION ABC clinic or training session as a patient, carer or Healthcare Professional

Exclusion Criteria:

* Unable to give informed consent
* Level of literacy precludes inclusion in questionnaire-based study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients invited to a MISSION ABC clinic, all Healthcare Professionals attending.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of clinic process measured through the collection of qualitative feedback. | up to 18 months
  Qualitative feedback forms collected at ever clinical encounter, qualitative interviews at 3 months post clinic and HCP focus groups will generate qualitative data. This will be evaluated cyclically to inform changes in the clinic structure.

SECONDARY OUTCOMES:
Number of changes in primary diagnosis or classification of disease severity resulting from a MISSION clinic appointment. | 18 months
  The number of new or changed diagnoses made as a result of a MISSION clinical encounter will be recorded.
Number of additional co-morbid medical conditions identified from a MISSION clinical encounter. | 18 months
  The number of co-morbid medical conditions identified by the medical team at a MISSION clinic will be recorded
Frequency of uptake and attendance at the enhanced asthma education programme ESMENA | 18 months
  The number of patients invited to attend ESMENA who accept the invitation will be recorded. Attendance rates over each 3 sessions will be recorded.
Changes in patients' perceived confidence in self-management before and after MISSION clinics and education sessions measured through questionnaire feedback | 18 months
  Patients will be asked to fill out a baseline questionnaire exploring their confidence in managing their disease and their health behaviours. They will be asked to rate confidence using a Liekrt scale that will be repeated at 3 and 6 months following their clinical or educational encounters.
Uptake and acceptability of HCP education through the MISSION process | 18 months
  The numbers and grade of HCP who attend MISSION clinics and dedicated education sessions will be recorded. 10% attendees will be asked to participate in focus group interviews which will explore their beliefs around the value and acceptability of these educational opportunities.
Number of patients where inhaler technique is improved at the first MISSION clinical encounter | 18 months
  Each patient will undergo an assessment of inhaler technique at their first appointment. Where education is required, it will be recorded if that intervention results in improvement.
Number of referrals to the smoking cessation service embedded in the MISSION clinics that results in a quit attempt | 18 months
  Data will be extracted from the GP record to indicate if a quit attempt is made
Any change in medication recorded | 18 months
  The number of new, changed or stopped prescriptions will be recorded.
Number of triggers on remote monitoring that can be managed remotely | 18 months
  The number of patients using the Message Dynamics or Clinitouch remote monitoring systems who trigger a positive response on symptoms or observations where they can be managed via a supported call rather than a GP attendance will be recorded. Any suspected delay in reporting disease deterioration due to the presence of the remote monitoring systems will also be recorded.
Number of additional secondary care referrals made as a result of the MISSION ABC process. | 18 months
  As a balancing measure, any secondary care referrals made will be recorded and additional costs to the healthcare system calculated.
Change in disease-specific symptom control questionnaires from baseline to 3 and 6 months | 6 months
  CAT or ACQ will be measured at baseline and then 3 and 6 months to assess changes in symptom control
Change in the productivity measure WPA from baseline to 3 and 6 months | 6 months
  Each patient will be asked to fill in the WPA at baseline, 3 and 6 months and the answers compared
Change in the patient activation measure from baseline to 3 and 6 months. | 6 months
  Each patient will be asked to fill in the PAM at baseline, 3 and 6 months and the answers compared
Changes in unscheduled health care usage per patient in the 12 months before and after MISSION ABC | 24 months
  For each patient the investigators will record their number of exacerbations, unscheduled GP visits, out-of-hours service calls, ED attendances and admissions in the 12 months before and 12 months after the MISSION clinic.
Acceptability of each innovation measured | 18 months
  MISSION ABC incorporates several innovative diagnosis and treatment solutions: Thorasys oscillometry, Flo-Tone devices, Airsonett laminar airflow, my mHealth online education, Message Dynamics Remote Monitoring, Clinitouch remote monitoring. For each device patients will be asked to give qualitative feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heiden E, Longstaff J, Chauhan MJA, DeVos R, Lanning E, Neville D, Jones TL, Begum S, Amos M, Mottershaw M, Micklam J, Holdsworth B, Rupani H, Brown T, Chauhan AJ; Mission ABC Collaborators. MISSION ABC: transforming respiratory care through one-stop multidisciplinary clinics - an observational study. BMJ Open. 2024 Jan 8;14(1):e078947. doi: 10.1136/bmjopen-2023-078947. PMID 38191248
- [Derived] Fox L, Heiden E, Chauhan MAJ, Longstaff JM, Balls L, De Vos R, Neville DM, Jones TL, Leung AW, Morrison L, Rupani H, Brown TP, Stores R, Chauhan AJ. Evaluation of telehealth support in an integrated respiratory clinic. NPJ Prim Care Respir Med. 2022 Nov 11;32(1):51. doi: 10.1038/s41533-022-00304-9. PMID 36369507